CLINICAL TRIAL: NCT05203549
Title: Consistency Between Treatment Responses in Patient-Derived Organoid (PDO) Models and Clinical Outcomes of Neoadjuvant Therapy, Conversion Therapy and Palliative Therapy in Gastric Cancer
Brief Title: Consistency Between Treatment Responses in PDO Models and Clinical Outcomes in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D1 Medical Technology (Shanghai) Co., Ltd, China (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D1med-GC1001
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A part of the tumor will be removed from the primary tumor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric cancer patients: Patients with gastric cancer will undergo tumor biopsy before receiving neoadjuvant therapy, conversion therapy, or palliative therapy
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor biopsy — Patients with gastric cancer will undergo tumor biopsy before receiving neoadjuvant therapy, conversion therapy, or palliative therapy

SUMMARY:
Gastric cancer is the fourth leading cause of cancer-related death worldwide. Accurate assessment of the clinical responses to current treatment regimens is key to improving the prognosis and prolonging the survival of patients. In this study, two hundred and fifty patients with gastric cancer who ought to receive neoadjuvant therapy, conversion therapy or palliative chemotherapy will be enrolled, and patient-derived organoids from their tumor biopsies will be used to test the sensitivity of chemotherapy drugs which mainly include 5-fluorouracil, irinotecan, oxaliplatin and paclitaxel.

DETAILED DESCRIPTION:
Two hundred and fifty stage II-IV gastric cancer patients who should receive neoadjuvant therapy, conversion therapy or palliative chemotherapy will be enrolled in this study. Baseline information of the enrolled patients including medical history, physical examination records and clinical examination records will be collected. Tumor material of those patients will be obtained from gastric endoscopic biopsies or surgical resection. Patient-derived organoids (PDOs) will be established and cultured from gastric cancer tumor specimens. PDOs will then be treated with drugs of the chemotherapeutic regimens for gastric cancer. Organoid size and growth will be monitored before and after the treatment, and dose-response curves will be generated. As for the assessment of clinical outcomes of patients, tumor regression grade (TRG) systems will be used to evaluate tumor histological responses, and treatment responses will also be assessed by biomedical imaging according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1). Consistency between treatment responses in PDO models and clinical outcomes of patients will be assessed by correlation analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 70 years old, no gender limit
2. The primary tumor is diagnosed as gastric adenocarcinoma (papillary, tubular, signet ring cell, poorly differentiated and mucinous adenocarcinoma) by endoscopic biopsy sampling and follow-up histopathological staining
3. The pre-operative staging includes: a) Stage IVa（cT4bNanyM0），resectable; b) Stage II-III（cT1-2N1-3M0、cT3-4aN0-3M0）, gastro-oesophageal junction (GEJ) cancer；c) Stage III（cT3-4aN1-3M0）, non-GEJ cancer, appropriate for neoadjuvant therapy
4. Stage IVb or locally unresectable late-stage gastric or GEJ cancer, previously never received chemotherapy
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
6. The function of major organs is normal, meeting the following criteria: a) routine blood tests (no blood transfusion in the past 14 days): HB≥90g/L；ANC ≥1.5×109/L；PLT ≥80×109/L；b）blood biochemical parameters: BIL <1.5-fold upper limit of normal (ULN)；ALT<2.5×ULN; AST<2.5×ULN；Crea≤1×ULN
7. Fresh tumor tissue biopsies are obtainable and the clinical information of the patients is complete
8. Patients have been informed and consented

Exclusion Criteria:

1. Previously received neoadjuvant therapy
2. Previously had other types of malignancy and received chemotherapy or radiotherapy
3. Previously had chicken pox, herpes zoster or other severe contagious diseases
4. Have severe active ulcer (gastrointestinal tract, skin, etc.) or have developed a high fever
5. Have a medical history of myocardial infarction, cerebral infarction, or pulmonary embolism
6. Have complications of gastric cancer (bleeding, perforation and obstruction etc.) and need emergency operation
7. Pregnant or lactating women
8. Have severe mental diseases
9. Allergic to chemotherapy drugs
10. Have metastatic brain cancer
11. Refuse to cooperate and to complete a treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred and fifty patients with gastric cancer who need to receive neoadjuvant therapy, conversion therapy or palliative chemotherapy are included in this study.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of patient-derived organoids | 2021.05 - 2023.12
  Patient-derived organoids (PDOs) will be established from gastric cancer tumor specimens and the rate of successful generation of gastric cancer organoids will be calculated.

SECONDARY OUTCOMES:
Correlation between results of the drug sensitivity tests in patient-derived organoid models and clinical outcomes | 2021.05 - 2023.12
  The results from drug sensitivity tests in patient-derived organoid models will be compared with clinical outcomes after neoadjuvant therapy, conversion therapy and palliative therapy, followed by correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No